CLINICAL TRIAL: NCT06877143
Title: Hypercaloric PEG Nutrition in ALS to Sustain Energy Homeostasis
Acronym: PEGASUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Albert Christian Ludolph, Prof., Prof. Dr., University of Ulm
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 387/23; PEGASUS V 1.0 (Other: Ulm University, GERMANY)
Record Dates: First submitted 2025-02-26; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: ALS; PEG; hypercaloric nutrition; energy deficit
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: randomized controlled double-blind study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Isocaloric nutrition via PEG (Other): Isocaloric nutrition (100% of individual calory requirement as determined by indirect calorimetry and physical activity questionnaire) applied via PEG
  Interventions: Dietary Supplement: 100% of individual calory requirement
- Group B: Hypercaloric nutrition via PEG (Experimental): Hypercaloric nutrition (120% of individual calory requirement as determined by indirect calorimetry and physical activity questionnaire) applied via PEG
  Interventions: Dietary Supplement: 120% of individual calory requirement

INTERVENTIONS:
Dietary Supplement: 100% of individual calory requirement — Patients receive any PEG nutrition containing the calory requirement as determined by indirect calorimetry, physical activity score and the randomized group.
  Arms: Group A: Isocaloric nutrition via PEG
Dietary Supplement: 120% of individual calory requirement — Patients receive any PEG nutrition containing the calory requirement as determined by indirect calorimetry, physical activity score and the randomized group.
  Arms: Group B: Hypercaloric nutrition via PEG

SUMMARY:
Weight loss is a known negative prognostic factor in amyotrophic lateral sclerosis (ALS). Over the last years, various interventional studies targeting the energy deficit in ALS yielded promising results; however,it is still unclear which kind of nutrition or nutritional supplement is most beneficial. Moreover, there is lack of evidence regarding interventions in patients with a PEG in later disease stages.In a pilot study conducted in 2013, it was demonstrated that body weight can be stabilized in ALS by applying either a fat-rich or carbohydrate-rich high-caloric food supplement. In 2014, Wills et al. conducted a placebo-controlled randomized controlled pilot study, which indicated that a carbohydrate-rich, hypercaloric diet, consisting in 125% of estimated energy requirements as determined by indirect calorimetry, in patients fed via percutaneous endoscopic gastrostomy was safe and well tolerated. Moreover, these patients showed longer survival than patients fed with a fat-rich, hypercaloric diet or an isocaloric diet . Hypercaloric, high-carbohydrate diet also showed beneficial effects on body weight and Body Mass Index . Although these results were promising, the low number of patients (n=24) was a severe limiting factor of this study. The aim of this study is to investigate the effect of a hypercaloric PEG nutrition, consisting of 120% of estimated calorie requierements, compared to an isocaloric nutrition. Individual energy requirement is determined by performing indirect calorimetry and activity questionnaire. The investigators hypothsize, that a hypercaloric PEG nutrition slows down disease progression as measured by neurofilament light chains (NfL) in serum after 6 months compared to placebo. Power calculation relies on the results of the lipids and calories for ALS (LIPCAL-ALS) study which tested the effect of an oral high-caloric fatty nutritional supplement in ALS. The study revealed that NfL serum values declined significantly in the intervention group while remaining stable in the placebo group over the course of the study. Assuming a similar effect size, we calculated that 76 patients had to be included in the current trial.

DETAILED DESCRIPTION:
Patients eligible for study participation will be randomized to one of two groups (hypercaloric or isocaloric diet) at baseline visit. Intervention or control diet will be administered as an add-on to standard therapy. Calory requirement will be individually determined by indirect calorimetry which measures resting energy expenditure (REE) and by collecting physical activity data. Indirect calorimetry is a non-invasive procedure which allows to calculate resting energy expenditure by measuring carbon dioxide and oxygen in the expired air using a canopy hood or a full-face mask. For both groups, a standard PEG nutrition featuring a balanced ratio of fat, carbohydrates, and protein according to human requirements will be used (e.g. Fresenius Fresubin® Energy Fibre/2250 Complete).

PEG nutrition used in this study (e.g. Fresenius Fresubin® Energy Fibre/2250 Complete) is routinely used in clinical practice for feeding of patients with ALS and PEG. It is known to be well tolerable and safe. In few cases of intolerance, this standard tube feeding may be switched to another product (e. g. HiPP Sondennahrung), but the amount of calories will not be changed.

In clinical routine, energy needs are usually estimated using the Harris-Benedict-formula, based on body weight, height, sex and age. However, this formula only provides approximate values. Therefore, in this study, indirect calorimetry is used to obtain precise values of energy needs. The German version of the International Physical Activity Questionnaire Short Last 7 Days Self-administered Format (IPAQ) is used for determining the physical activity level. The total energy requirement is calculated by adding the resting energy expenditure and the activity-related calorie requirement.

In the control group, 100% of the estimated calorie requirement is administered with the goal of covering energy needs and stabilizing body weight. The hypercaloric diet in the intervention group consists in 120% of the calorie requirement determined by indirect calorimetry. Resting energy expenditure in ALS patients is 14% higher than in a healthy control cohort. We assume that activity-related energy expenditure is increased similarly. Therefore, the hypercaloric diet consisting in 120% of calorie requirement aims to cover these additional energy needs. Similarly, a recent study in patients with PEG used 125% of calorie requirement.

ELIGIBILITY:
Inclusion Criteria:

* Possible, probable (clinically or laboratory) or definite ALS according to the revised version of the El Escorial World Federation of Neurology criteria 1
* Loss of ALS functional rating scale revised (ALSFRS-R) of ≥ 0.33 points per month since onset (first paresis) based on the formula: (48 - Score at Screening Visit) / (Months between Onset and Screening Visit)
* Nutrition via PEG
* Age ≥18 years
* Intake of a stable dose of riluzole for at least 4 weeks, or no riluzole
* Capable of thoroughly understanding all information given and giving full informed consent according to GCP

Exclusion Criteria:

* Previous participation in another interventional study within the preceding 4 weeks
* Absence of adequate social support and cooperation, or personal motivation (in the judgment of the investigator) to complete the study satisfactorily
* Pregnancy or breast-feeding females
* Evidence of a major psychiatric disorder or clinically evident dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Neurofilament light chain (NfL) in serum | 6 months
  Change of neurofilament light chain (NfL) concentration in serum after 6 months compared to baseline. The change will be measured as individual NfL slope from baseline to 6 months (change per month).

SECONDARY OUTCOMES:
Survival | 6 months
  time to death or tracheostomy
ALS functional rating scale revised (ALSFRS-R) | 6 months
  Amyotrophic Lateral Sclerosis Functional Rating Scale Revised (ALSFRS-R) score, measured as individual slope (loss of points per month)
Body mass index (BMI) | 6 months
  Body Mass Index (BMI), weight (in kg) and height (in m) will be combined to report BMI in kg/m^2
Slow vital capacity | 6 months
  Slow vital capacity (sVC)
Resting energy expenditure (REE) | 6 months
  Resting Energy Expenditure (REE), measured by indirect calorimetry
Individual Quality of Life | 6 months
  Individual Quality of Life, measured by the Euro Quality of Life (EQ-5D-5L) questionnaire
Appetite | 6 months
  Appetite, measured by the Council of Appetite Questionnaire (CNAQ)
Eating habits | 6 months
  Eating Habits, evaluated by the Ulm Nutrition Questionnaire (UNQ; see LIPCAL study)
Adverse Events | 6 months
  Terms and frequencies of adverse eves (AEs) and serious adverse events (SAEs)
Fatt mass | 6 months
  Fat mass (% of total body mass), measured by bioelectrical impedance analysis (BIA)
Total Body Water | 6 months
  total body water (% of total body mass), measured by bioelectrical impedance analysis (BIA)
Muscle Mass | 6 months
  muscle mass (% of total body mass) measured by bioelectrical impedance analysis (BIA)
Fat Free Mass | 6 months
  fat free mass (% of total body mass), measured by bioelectrical impedance analysis (BIA)
Body Cell Mass | 6 months
  body cell mass (% of total body mass), measured by bioelectrical impedance analysis (BIA)
Extracellular Mass | 6 months
  extracellular mass (% of total body mass), measured by bioelectrical impedance analysis (BIA)
Lean Body Mass | 6 months
  lean body mass (% of total body mass), measured by bioelectrical impedance analysis (BIA)
Beta Hydroxybutyrate | 6 months
  Beta Hydroxybutyrate serum levels
Acetoacetate | 6 months
  Acetoacetate serum levels
Acetone | 6 months
  Acetone concentration in urine
Lipid metabolism | 6 months
  Cholesterol serum levels
Lipid metabolism | 6 months
  High-density-lipoprotein (HDL) serum levels
Lipid metabolism | 6 months
  Low-density-lipoprotein (HDL) serum levels

CONTACTS AND LOCATIONS:
Overall Officials: Christine Herrmann, Dr., Principal Investigator — University of Ulm
Locations (1):
- Ulm Universita, Department of Neurology, Ulm, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data after de-identification as well as the study protocol will be available. Data will be available beginning 3 months and ending 5 years following article publication. Data will be shared with researchers who provide a methodologically sound proposal. Data will be shared for analyses to achieve the aims provided in the approved proposal. Proposals should be directed to christine.herrmann@uni-ulm.de; to gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol
Time Frame: 3 months to 5 years following article publication
Access Criteria: Data will be shard for analyses to achieve the aims provided in the approved proposal. Proposals should be directed to christine.herrmann@uni-ulm.de; to gain access, data requestors will need to sign a data access agreement.
URL: https://www.uniklinik-ulm.de/neurologie.html

REFERENCES:
- See also: Desport JC, Preux PM, Truong TC, Vallat JM, Sautereau D, Couratier P. Nutritional status is a prognostic factor for survival in ALS patients. Neurology 1999; 53(5): 1059-63. — https://pubmed.ncbi.nlm.nih.gov/10496266/
- See also: Dupuis L, Oudart H, Rene F, Gonzalez de Aguilar JL, Loeffler JP. Evidence for defective energy homeostasis in amyotrophic lateral sclerosis: benefit of a high-energy diet in a transgenic mouse model. Proc Natl Acad Sci U S A 2004; 101(30): 11159-64. — https://pubmed.ncbi.nlm.nih.gov/15263088/
- See also: Dupuis L, Pradat PF, Ludolph AC, Loeffler JP. Energy metabolism in amyotrophic lateral sclerosis. Lancet Neurol 2011; 10(1): 75-82. — https://pubmed.ncbi.nlm.nih.gov/21035400/
- See also: Fayemendy P, Marin B, Labrunie A, et al. Hypermetabolism is a reality in amyotrophic lateral sclerosis compared to healthy subjects. J Neurol Sci 2021; 420(117257): 3. — https://pubmed.ncbi.nlm.nih.gov/33290920/
- See also: Dorst J, Cypionka J, Ludolph AC. High-caloric food supplements in the treatment of amyotrophic lateral sclerosis: A prospective interventional study. Amyotroph Lateral Scler Frontotemporal Degener 2013; 14(7-8): 533-6. — https://pubmed.ncbi.nlm.nih.gov/23944684/
- See also: Ludolph AC, Dorst J, Dreyhaupt J, et al. Effect of high-caloric nutrition on survival in amyotrophic lateral sclerosis. Ann Neurol 2019; 17(10): 25661. — https://pubmed.ncbi.nlm.nih.gov/31849093/
- See also: Dorst J, Schuster J, Dreyhaupt J, et al. Effect of high-caloric nutrition on serum neurofilament light chain levels in amyotrophic lateral sclerosis. J Neurol Neurosurg Psychiatry 2020; 91(9): 1007-9. — https://pubmed.ncbi.nlm.nih.gov/32788256/
- See also: Steinacker P, Huss A, Mayer B, et al. Diagnostic and prognostic significance of neurofilament light chain NF-L, but not progranulin and S100B, in the course of amyotrophic lateral sclerosis: Data from the German MND-net. Amyotroph Lateral Scler Frontotem — https://pubmed.ncbi.nlm.nih.gov/27819158/
- See also: Wills AM, Hubbard J, Macklin EA, et al. Hypercaloric enteral nutrition in patients with amyotrophic lateral sclerosis: a randomised, double-blind, placebo-controlled phase 2 trial. Lancet 2014; 383(9934): 2065-72. — https://pubmed.ncbi.nlm.nih.gov/24582471/
- See also: Dorst J, Dupuis L, Petri S, et al. Percutaneous endoscopic gastrostomy in amyotrophic lateral sclerosis: a prospective observational study. J Neurol 2015. — https://pubmed.ncbi.nlm.nih.gov/25618254/
- See also: Wang S, Yuan T, Yang H, Zhou X, Cao J. Effect of complete high-caloric nutrition on the nutritional status and survival rate of amyotrophic lateral sclerosis patients after gastrostomy. American journal of translational research 2022; 14(11): 7842-51. — https://pubmed.ncbi.nlm.nih.gov/36505314/
- See also: Craig CL, Marshall AL, Sjöström M, et al. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc 2003; 35(8): 1381-95. — https://pubmed.ncbi.nlm.nih.gov/12900694/